CLINICAL TRIAL: NCT07072832
Title: Shelf Acetabuloplasty With 3D Printed Implants as a New Treatment for Symptomatic Adult Hip Dysplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Replasia BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: version 1.2 d.d 28-11-2024
Record Dates: First submitted 2025-06-18; First posted 2025-07-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Hip Dysplasia
Keywords: Dysplasia; Hip; Adult; Preservation; Shelf
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment group (Experimental): Consisting of two sequential cohorts. Five patients first treated in safety cohort, five patients after in performance cohort.
  Interventions: Device: 3D-Shelf

INTERVENTIONS:
Device: 3D-Shelf — Treatment of hip dysplasia using novel 3D printed 3D-Shelf device.

SUMMARY:
Hip dysplasia is a common orthopedic condition, defined as an abnormality in the shape, size and orientation of the femoral head, acetabulum or both. The most frequent presentation of hip dysplasia is the maldevelopment of the acetabulum, resulting in insufficient superior coverage of the femoral head, defined as a lateral center-edge angle (Wiberg) of less than 20 degrees. Patients suffer from groin pain, an abnormal gait, decreased strength, and an increased rate of degenerative hip disease.

The possible treatments affecting the shape of the acetabulum once the patient reaches adolescence are all surgical. The PAO is regarded as the current gold standard in the treatment of symptomatic adult hip dysplasia. The 3-dimensional orientation of the acetabulum is changed with the use of 3 osteotomies around the acetabulum and a refixation in the obtained position. However, the PAO is a difficult operation and is associated with a large number of major complications (up to 37%), and the surgery is associated with a long rehabilitation period.

Hence, a strong unmet need exists for an effective but less invasive solution that enhances the quality of life of adult hip dysplasia patients. The treatment gap can be filled with a 3-dimensional (3D) shelf procedure. This custom-made implant (called the 3D-Shelf implant) was developed with the goal to be more predictable in terms of containment and fit than the old autologous shelf-acetabuloplasty, and less invasive and easier to perform than the PAO.

This study aims to study the safety and evaluate the early performance in terms of the clinical outcomes after implantation of the 3D-Shelf implant in patients with adult hip dysplasia, to show that the 3D-Shelf procedure is safe, has lower complication rates, and shows no inferiority in clinical outcomes compared to the current treatment of a peri-acetabular osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* Hip dysplasia based on AP x-ray with a LCEA of <25°
* Groin pain and/or gait abnormalities, with no other explanatory hip pathology
* Aged at least 18 years and maximal 45 years at time of surgery (indicated age for PAO(19))
* Willing to comply with the study visit schedule during 12 month follow-up
* Able and willing to provide informed consent

Exclusion Criteria:

* Previous acetabular surgery >10yr of age
* Signs of osteoarthritis on x-ray (Tonnis classification >1),
* Body mass index of more than 35
* Large labral tears visible on non-contrast MRI
* Pre-consultation known titanium allergy
* Pre-consultation known medical histories of diseases that per the investigator possibly affect the outcome: neuromuscular disease affecting the stability of the hip, diseases affecting bone ingrowth and fixation strength of the implant like rheumatoid arthritis and metabolic bone diseases, e.g. osteomalacie, osteoporosis, hyperparathyroidism, hypercalcemia.
* Pre-consultation known pregnant women or women who are planning to become pregnant during the duration of the study.
* Part of vulnerable population (e.g. Mentally disabled with cognitive impairment or mental disease)
* Currently participating in another investigational clinical trial.
* Unable to provide informed consent (e.g. insufficient language skills)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
PROMs | from baseline (pre-surgery), 3 months, 6 months and 12 months.
  Performance and safety will be evaluated using patient-reported outcome measures, specifically the International Hip Outcome Tool (iHOT-33), which assesses health-related quality of life in young, active patients with hip disorders. Scores range from 0 to 100, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Implant position | 24 hours after surgery and 12 months after surgery
  Evaluation of the implant position using CT
Recovery time | From 3 months, 6 months and 12 months
  Patient recovery will be evaluated through a combination of patient-reported and clinical outcomes. Patient-reported outcomes include the International Hip Outcome Tool (iHOT-33), which ranges from 0 to 100 with higher scores indicating better function and quality of life, and the EQ-5D. Clinical assessment will include evaluation of hip range of motion and return to normal function as judged by the investigator.
Surgical risks | From surgery to end of follow-up (12 months)
  Evaluation of surgical risks will include monitoring and documentation of surgery-related adverse events and any deviations from the planned surgical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Ziekenhuis, Geldrop, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
To be determined.